CLINICAL TRIAL: NCT00143169
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study Of Morphine-Sparing Effect And Safety Of Parecoxib Administered Intravenously For The Treatment Of Postoperative Pain Following Orthopedic Or Gynecological Surgery
Brief Title: Morphine-Sparing Effect And Safety Of Parecoxib Administered Intravenously For The Treatment Of Postoperative Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A3481004
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2008-04-15 (Estimated); Status verified 2005-11

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — parecoxib

INTERVENTIONS:
Drug: Parecoxib and placebo

SUMMARY:
To validate the morphine-sparing effect and safety of parecoxib administered intravenously for the treatment of Chinese subjects with postoperative pain following gynecological or orthopedic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergo gynecological or orthopedic surgery under epidural anesthesia

Exclusion Criteria:

* A previous history of intolerance or hypersensitivity to any NSAID, cyclooxygenase-2 selective inhibitors, sulphonamides, or any of the excipients of parecoxib.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220
Dates: Start 2004-09; Study Completion 2005-06

PRIMARY OUTCOMES:
To validate the morphine-sparing effect of parecoxib administered intravenously for the treatment of Chinese subjects with postoperative pain following gynecological or orthopedic surgery.

SECONDARY OUTCOMES:
To validate safety of parecoxib administered intravenously for the treatment of Chinese subjects with postoperative pain following gynecological or orthopedic surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- China (5):
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Qingdao, Shandong
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Shanghai